CLINICAL TRIAL: NCT07209644
Title: Serum Catestatin in Systemic Sclerosis: Relations to Cardiovascular Involvement and Microvascular Alterations
Brief Title: Catestatin as a Novel Biomarker for Cardiovascular and Microvascular Involvement in Systemic Sclerosis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa awwad abdoh radwan, resident at the Rheumatology, Rehabilitation and Physical Medicine department, Assiut University
Other Study IDs: Serum Catestatin
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Systemic Sclerosis
Keywords: Systemic sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Systemic Sclerosis Arm: Patients with systemic sclerosis (n=35), assessed for disease activity, catestatin levels, cardiovascular involvement, and microvascular changes.
- Control Arm: Healthy controls (n=35), evaluated for serum catestatin levels to provide a baseline reference.

SUMMARY:
This study investigates the relationship between serum catestatin levels and systemic sclerosis (SSc), with a focus on cardiovascular involvement and microvascular alterations, to determine catestatin's potential as a biomarker of disease activity and severity.

DETAILED DESCRIPTION:
Systemic sclerosis is a chronic autoimmune disease characterized by fibrosis, autoimmunity, and vasculopathy, with cardiovascular complications accounting for a significant proportion of morbidity and mortality. Despite advances in diagnostic tools, early identification of high-risk patients remains challenging. Catestatin, a peptide derived from chromogranin A, has recently gained attention as a biomarker with regulatory roles in cardiovascular physiology, including hypertension, endothelial function, and vascular remodeling. This cross-sectional study will assess serum catestatin levels in patients with SSc compared with healthy controls. It aims to correlate these levels with disease activity indices, cardiovascular involvement (using echocardiography, ECG, and blood pressure monitoring), and microvascular abnormalities identified via nailfold capillaroscopy. Findings from this study may establish catestatin as a promising biomarker, paving the way for improved management and cardiovascular risk stratification in SSc patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with systemic sclerosis according to 2013 ACR-EULAR classification criteria.

Age >18 years.

Exclusion Criteria:

* Other autoimmune disorders.

Cardiovascular conditions not linked to systemic sclerosis.

Comorbidities affecting catestatin metabolism (e.g., diabetes, chronic kidney disease, obesity).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will include 35 patients diagnosed with systemic sclerosis according to the 2013 ACR-EULAR classification criteria and 35 age- and sex-matched healthy controls without autoimmune or cardiovascular diseases. Patients must be over 18 years old, and both genders will be included. Controls will be recruited from hospital staff and volunteers. Exclusion criteria eliminate any confounding factors affecting serum catestatin, including other autoimmune diseases, comorbid cardiovascular conditions unrelated to SSc, diabetes, chronic kidney disease, and obesity.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
change in level of serum catestatin concentration in systemic sclerosis patients compared with healthy controls. | baseline
  Quantification of serum catestatin levels using ELISA, directly compared between the two study groups.